CLINICAL TRIAL: NCT05148247
Title: Evaluation of The Perceive, Recall, Plan and Perform Intervention for Persons With Cognitive Impairments After Brain Injuries in Community Rehabilitation: Single Case Experimental Study
Brief Title: Occupational Therapy and Cognitive Challenges After Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Østre Toten Municipality (Unknown); Skien Municipality (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REK 215391
Record Dates: First submitted 2021-10-29; First posted 2021-12-08 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Brain Injuries; Cognitive Impairment
Keywords: Task Performance; Occupational Therapy; Community Health Services; Elderly; The Perceive, Recall, Plan and Perform System; Rehabilitation
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction; Neuroaxonal Dystrophies

STUDY DESIGN:
Intervention Model Description: Single-Case Experimental Designs with Multiple baselines across participants. At least five data collection points within 4 phases (= at least 20 data points) for each participant (= one tier), and a minimum of three participants (= one sample), is recommended to meet design quality standards. The 'Number of Arms' will in this tradition mean one tier. Data for at least 2 samples will be collected, each of 3 tiers.
Masking Description: Participants are randomized to three different baseline-lengths in each tier, that serve as control data in this design. Blinding is not possible for the conducting OT, but an independent PRPP-trained OT assesses 20 % of the PRPP stage 1 and 2 measurements from each phase by videotaping the assessment situations. The tapes will be presented blinded and randomly for this second and blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PRPP Intervention (Experimental): This baseline phase will be 3, 5 or 7 days, and intervention phase starts immediately after baseline with 45-60 minutes PRPP Intervention 3 times a week for 3 weeks.
  Interventions: Behavioral: The Perceive, Recall, Plan and Perform System of Intervention

INTERVENTIONS:
Behavioral: The Perceive, Recall, Plan and Perform System of Intervention — The aim of the PRPP intervention is to enhance mastery in performance of needed or desired occupations, and extend traditional task training. Systematic instructions to support the clients' cognitive capacity to think about doing in different tasks and contexts are given by the OT, based on the results of PRPP Assessment stage 2. Further, the OT uses graded verbal, visual or physical prompts and cues directly during the participants task performance, progressing from content-free meta-prompts 'Stop' to alert the participant to process information required for the task, and for errorless learning. Then the OT prompt 'sense/attend, think and do', to more specific behavioural prompts selected by the therapist based on the components from the PRPP Assessment stage 2. At best the skills are generalized throughout all everyday activities, and the OTs' role as a cognitive mediator fades as the person internalize the strategies.
  Other Names: PRPP

SUMMARY:
Background: There is a need for standardized interventions in community rehabilitation that can improve everyday task performance for older adults with cognitive challenges after acquired brain injury. Older adults are often excluded from research due to strict inclusion criteria. It is critical for a sustainable health service system that these patients are empowered and reach their maximum level of independence. The Perceive, Recall, Plan and Perform System (PRPP) of Intervention can be applied by Occupational Therapists (OT) for clients with cognitive challenges to enhance mastery of needed or desired everyday tasks. There is no current evidence for the effectiveness of this intervention for this population.

Purpose: A clinical trial to investigate the effectiveness of the PRPP intervention for older persons with cognitive impairments after brain injury in the context of community-based rehabilitation.

Method: In PRPP intervention the OT uses systematically instructions in task training to support a client to use cognitive strategies efficiently. The everyday tasks used for training should be valued by the participant and useful in their rehabilitation. The tasks could include different parts of morning routines, simple or complex meal planning or preparation, use of cell phone, leisure activities, or other household and community activities. At best the skills are generalized throughout all everyday activities, and the OTs' role as a cognitive mediator fades as participants internalize the strategies. The participants receive PRPP intervention 3 times a week for 3 weeks, every session last for 45-60 minutes.

The participants' task mastery and cognitive strategy use will be measured at least 5 times in each phase: baseline, intervention, after the intervention, and 4 weeks after the discharge from rehabilitation. The measurement scores at baseline act controls and are therefore compared with the other phases for the same participant. The same procedure will be repeated for the other participants, but then with a staggered intervention phase. A staggered intervention phase acts as a control between participants and allows to see if changes occur only when the intervention is introduced.

Implications for practice: The investigators assume that this systematic intervention will improve everyday task performance, and will in turn contribute to empowerment and independence of older adults with cognitive challenges after brain injuries.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the health centres in the two municipalities
* Acquired brain injury
* Mastery under 85% of PRPP Assessment stage 1

Exclusion Criteria:

* An already diagnosed dementia or progressive brain disorder
* Congenital brain injury or neurological developmental disorder
* Not able to understand or hear instructions, due to foreign language, severe hearing loss or severe arousal problems
* Physical disabilities that hinder performance of most daily activities.
* If a participant show mastery above 85% of PRPP Assessment stage 1, the participant either need to be assessed in more taxonomic difficult activities or will be excluded with 'no cognitive challenges in occupational performance'.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Change in task performance | Is measured at 5 points in each of the 4 phases; in the baseline phase of the 3, 5 or 7 first days after referral to OT, during 3 weeks of intervention phase, the 2 following days as post-intervention, and 4 weeks after discharge to home.
  Five everyday tasks will be target behavior, and each will be divided into a series of significant steps and measured in percentage mastery of the steps according to "The Perceive, Recall, Plan and Perform Assessment stage 1" as a functional measure. The highest score is 100% mastery of the steps, and the lowest is 0%, where none of the steps have appropriate mastery. With a score above 85% the participant is considered as independent, but with minor errors in performance.

SECONDARY OUTCOMES:
Change in cognitive strategy application | Is measured at 5 points in each of the 4 phases; in the baseline phase of the 3, 5 or 7 first days after referral to OT, during 3 weeks of intervention phase, the 2 following days as post-intervention, and 4 weeks after discharge to home.
  "The Perceive, Recall, Plan and Perform Assessment stage 2" (PRPP) is used to measure the effectiveness of 34 observable cognitive strategy application behaviours in the everyday task performance.The PRPP Assessment stage 2 is criterion-referenced and evaluated in a three-point scale: (3) effective task performance, (2) questionable or (1) not effective. An effective performance in all the observable strategies will give a score of 102 points and with the lowest outcome of 34 points if all the cognitive strategy applications are not effective. For the therapist it will be even more valuable to notice which of the cognitive strategies that are not effective, as a foundation for the intervention.

OTHER OUTCOMES:
Change in the Barthel Index | Is measured all together three times, once in the baseline phase of 3, 5 or 7 days, the 2 following days after 3 weeks of the intervention phase in the post-intervention phase and after 4 weeks after discharge in a follow-up phase.
  The Barthel Index assess functional outcomes to measure independency in daily activities and will serve as generalization measures for the target behavior. The Barthel Index quantify the participants' performance in 10 activities of daily life, where the participants can be scored for 0, 5 or 10 points, with the highest score of 100 is the highest value and a score over 95 consider that the participant is independent in personal daily activities. A score of 0 is the lowest value and worse outcome.
Change in the Goal Attainment Scale | Is measured all together three times, once in the baseline phase of 3, 5 or 7 days, the 2 following days after 3 weeks of the intervention phase in the post-intervention phase and after 4 weeks after discharge in a follow-up phase.
  The Goal Attainment Scale is a method of quantifying the extent to which patient's individual goals are achieved in the course of intervention. The scores goes from -2, -1, 0, +1 and +2. The score of 0 is the baseline value, and better outcome is the scores of +1 and +2, whereas worse outcome is the -1 and -2 scores.

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Vifladt, Study Chair — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Østre Toten Municipality, Department of Physio- and Occupational Therapy, Lena
  - Skien Municipality, Department of Rehabilitation and Palliative Care, Skien

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Plan: The results of this project will be shared in scientific journals and clinical and scientific conferences.
  The research data will be used by the Project Manager, the PhD Candidate and students supervised by them until five years after the project ends (probably year 2029). After that, any data will be deidentified, and personal information will be deleted.
  Regarding the approval from the Regional Ethics Committee (REC, project number 215391) and the participant consent, data sharing with other research groups is not prepared for and planned. However, anonymized raw data generated with PRPP stages 1 and 2, The Goal Attainment Scaling and The Barthel Index are available upon reasonable request and can be used for purposes mentioned in the REC approval and participant consent.
  The data are in Norwegian, and a translation is not planned.
Supporting Information: Study Protocol, ICF
Time Frame: See plan description.
Access Criteria: Upon reasonable request to the Project Manager Dr. Linda Stigen.

REFERENCES:
- [Background] Porcino AJ, Shamseer L, Chan AW, Kravitz RL, Orkin A, Punja S, Ravaud P, Schmid CH, Vohra S; SPENT group. SPIRIT extension and elaboration for n-of-1 trials: SPENT 2019 checklist. BMJ. 2020 Feb 27;368:m122. doi: 10.1136/bmj.m122. No abstract available. PMID 32107202
- [Background] Tate RL, Perdices M, Rosenkoetter U, Shadish W, Vohra S, Barlow DH, Horner R, Kazdin A, Kratochwill T, McDonald S, Sampson M, Shamseer L, Togher L, Albin R, Backman C, Douglas J, Evans JJ, Gast D, Manolov R, Mitchell G, Nickels L, Nikles J, Ownsworth T, Rose M, Schmid CH, Wilson B. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) 2016 Statement. J Clin Epidemiol. 2016 May;73:142-52. doi: 10.1016/j.jclinepi.2016.04.006. Epub 2016 Apr 19. PMID 27101888
- [Derived] Lindstad MO, Obstfelder AU, Sveen U, Stigen L. Evaluating the PRPP Intervention for individuals with brain injury at local inpatient rehabilitation facilities: multiple baseline designs. Neuropsychol Rehabil. 2025 Nov 21:1-28. doi: 10.1080/09602011.2025.2590092. Online ahead of print. PMID 41270188
- [Derived] Lindstad MO, Obstfelder A, Sveen U, Stigen L. Effectiveness of the PRPP Intervention after brain injury in home-based rehabilitation: Single-case experimental designs with multiple baselines. Scand J Occup Ther. 2025 Jan;32(1):2444591. doi: 10.1080/11038128.2024.2444591. Epub 2025 Jan 2. PMID 39744963
- [Derived] Lindstad MO, Obstfelder AU, Sveen U, Stigen L. Feasibility of the Perceive, Recall, Plan and Perform system of intervention for persons with brain injury in community-based rehabilitation: a pilot for a multiple-baseline design study. BMJ Open. 2023 Jun 28;13(6):e067593. doi: 10.1136/bmjopen-2022-067593. PMID 37380207
- [Derived] Lindstad MO, Obstfelder AU, Sveen U, Stigen L. Effectiveness of the Perceive, Recall, Plan and Perform intervention for persons with brain injury in community-based rehabilitation: protocol for a single-case experimental design with multiple baselines. BMJ Open. 2022 Oct 5;12(10):e060206. doi: 10.1136/bmjopen-2021-060206. PMID 36198473